CLINICAL TRIAL: NCT02468362
Title: Long Term Outcomes After Laparoscopic Intersphincteric Resection With Total Mesorectal Excision for Low Rectal Cancer: a Double Blind Randomized Clinical Trial
Brief Title: Long Term Outcomes After Laparoscopic Intersphincteric Resection With Total Mesorectal Excision for Low Rectal Cancer.
Acronym: ISR-TME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Mohammad Ali ElDamshety, surgical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISR-TME
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Low Rectal Cancer
Keywords: Intersphincteric resection; laparoscopic rectal rescetion; total mesorectal excsison

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Laparoscopic group (Active Comparator)
  Interventions: Procedure: laparoscopic intersphincteric resection
- Open group (Active Comparator)
  Interventions: Procedure: open intersphincteric resection

INTERVENTIONS:
Procedure: laparoscopic intersphincteric resection — laparoscopic intersphincteric resection for low rectal cancer
  Arms: Laparoscopic group
Procedure: open intersphincteric resection
  Arms: Open group

SUMMARY:
Through a double blinded study, patients with low rectal cancer will be randomized into two equal groups to compare between the 5 year disease free survival as a primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Low rectal cancer below 5 cm from the anal verge
* Fit for laparoscopic total mesorectal excsion
* T2, T3 rectal cancer
* No distant metstasis

Exclusion Criteria:

* T1, AND T4
* Distant metastasis
* Tumor infiltrating the dentate line
* unwilling to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Disease Free survival | 5 years

SECONDARY OUTCOMES:
Local recurrence | 5 years
Distant metstasis | 5 years
5 year survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Osama Eldamshety, PhD, MD, Principal Investigator — Oncology centre of mansoura university; Sherif Kotb, PhD, MD, Principal Investigator — Oncology centre of mansoura university; Nazem Shams, PhD, MD, Principal Investigator — Oncology centre of mansoura university; Ashraf Khater, Phd, MD, Principal Investigator — Oncology centre of mansoura university